CLINICAL TRIAL: NCT06326710
Title: The 'Outdoor Rehab-Fit' App-based Physical Activity Education Intervention for Frail Older Adults in Hong Kong: a Feasibility Pilot Randomized Controlled Trial Study Protocol
Brief Title: The 'Outdoor Rehab-Fit' App-based Physical Activity Education Intervention for Frail Older Adults in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LEE Lok Chun Janet, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P0045122
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-04

CONDITIONS: Physical Inactivity; Frailty
MeSH Terms: conditions — Sedentary Behavior; Frailty | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mHealth Group (Experimental): This arm of participants will be receiving 4 sessions of face-to-face or online delivered mHealth intervention.
  Interventions: Behavioral: mHealth
- Control Group (Active Comparator): This arm of participants will be receiving 4 sessions of face-to-face or online exercise delivered health talks.
  Interventions: Behavioral: Health Talk

INTERVENTIONS:
Behavioral: mHealth — Participants receive 4 sessions of face-to-face or online delivered workshop on how to use the mobile app "Outdoor Rehab-Fit" to support their daily PA level. In addition to the workshop, participants have to go to public parks to practice what they have learnt from the mobile app.
  Arms: mHealth Group
Behavioral: Health Talk — Participants receive 4 sessions of face-to-face or online delivered health talks on the benefits different types of modified exercises for frail older adults (chair yoga, seated eight-section brocades, Otago and seated multi-component exercise). Each talk has an experiential session.
  Arms: Control Group

SUMMARY:
In recent years, research teams around the world have developed interventions to educate older adults to use outdoor exercise facilities (OEFs) to improve health outcomes like strength, balance, mobility, PA level, and weight. These interventions employed trainers or therapists to instruct, and monitor exercise training for older adults using the public accessible OEFs. Apart from therapist or trainer-led intervention, an Australian research team developed a mobile application, and social support strategies to help participants to use OEFs to enhance their aerobic and resistance-based PA.

A recent local in-depth qualitative study discovered that OEFs in Hong Kong attracted frailer older adults (i.e., those who recovered from a major illness or who has chronic diseases), and their caregivers to use OEFs to support and maintain their daily PA behavior. Some used OEFs to complement their formal rehabilitation sessions. It appears that OEFs in Hong Kong serves as an important health maintenance space for frailer older adults in the city to "age in place", yet educational training related to OEFs has been lacking over the years. Signage besides the exercise equipment has been the only education material for users over the years.

A mobile app-based physical activity education intervention will be developed for frail old adults in Hong Kong. The intervention has two components: (1) mobile app; and (2) face-to-face group session that teaches the how to use correctly and safely use OEF in public parks to maintain PA habits.

The main objective of this study is to evaluate the feasibility, acceptability, and pilot effectiveness of the 'Outdoor Rehab-Fit' App-based physical activity education intervention. Primary outcomes include recruitment rate, retention rate, attrition rate, attendance, perceived usefulness of the app. Secondary outcomes include exercise self-efficacy, mental well-being, physical activity level.

This study adopts a mixed-method design with quantitative and qualitative method. This study is a pilot randomized controlled trial, running for 4 months evaluating of the effectiveness of the mHealth intervention. 40 frail older adults will be randomized into (i) mHealth group or (ii) control group.

Quantitative analysis will be adopted to investigate the effectiveness of the 'Outdoor Rehab-Fit' App-based physical activity education intervention on the health outcomes of frail older adults. The qualitative component will consist of semi-structure interviews with the frail older adults to understand the acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling men or women aged 55 years or over
* meeting at least one items of the FRAIL scale
* passing the Physical Activity Readiness- Questionnaire
* owning a smart phone for daily use
* signing the informed consent documents

Exclusion Criteria:

* older adult participants who achieved adequate level of daily physical activity, as defined as engaging in moderate-to-vigorous intensity physical activity for at least 150 minutes per week
* scoring 0 or 5 in the FRAIL scale

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome: Recruitment rate | Baseline
  Will be assessed by study record e.g., attendance log in recruitment seminar. It is calculated based on the percentage of who signed up for the study and the total number of approached participants.
Feasibility outcome: Intervention completion rate | Month 1
  Will be assessed by a self-invented record form. It is calculated based on the percentage of completion of all intervention components (Including workshop attendance, app usage and outdoor practice).
Feasibility outcome: Attrition rate | Month 1
  Will be assessed by study record. It indicates the rate at which participants dropped out or discontinued their participation in the study.
Feasibility outcome: Attendance | Month 1
  Will be assessed by study record (e.g., attendance log). It is the percentage of sessions attended over all the offered sessions.
Acceptability outcome: Perceived Usefulness on Outdoor Rehab-Fit App | Month 1
  Will be assessed by self-invented questionnaire. It measures participant's perceptions of the app's usefulness. The questionnaire consists of 3 domains.Overall score ranges from 20 to 100. Higher score indicates higher perceived usefulness.
Acceptability outcome: Participants' views about the barriers and facilitation of the mHealth program | Month 1
  Will be assessed by semi-structured interview guide.

SECONDARY OUTCOMES:
Change in Physical activity level (Objective) at 1 month and 3 months | Baseline, Month 1, Month 3
  ActiGraphs will be used to collect objective data on moderate-to-vigorous intensity physical activity. It is validated wrist-worn tri-axial accelerometers capturing motion on three axes: vertical (Y), horizontal right-left (X), and horizontal front-back axis at a sampling frequency of 30hz.
Change in Physical activity level (Subjective) at 1 month and 3 months | Baseline, Month 1, Month 3
  Rapid Assessment of Physical Activity Scale will be used to measure physical activity level. The scale is a 9-item questionnaire that uses a yes-or-no response format. It covers the range of PA levels, from sedentary to regular vigorous PA (RAPA1), as well as strength training and flexibility (RAPA2). A RAPA1 score less than 6 means sub-optimal and is used as a benchmark for not meeting the standard recommendations for physical activity. A RAPA2 score less than 3 is considered as suboptimal, meaning inadequate attainment of anaerobic PA.
Change in Exercise self-efficacy at 1 month and 3 months | Baseline, Month 1, Month 3
  The Chinese version Exercise self-efficacy will be used to examine the degree of an individual's confidence in exercising regularly. It consisted of nine items rated on an 11-point Likert scale, where '0' represents 'not confident' and '10' represents 'very confident'. Answers from the nine questions were averaged to a score ranged from 0 to 10, with higher scores corresponding to higher confidence in performing exercise and higher exercise self-efficacy.
Change in Mental well-being at 1 month and 3 months | Baseline, Month 1, Month 3
  The Chinese version of the seven-item short Warwick-Edinburgh Mental Well-Being Scale will be used to measure mental well-bing. The questions, which covered both hedonic and eudemonic aspects, were rated on a 5-point Likert scale, where '1' indicated 'none of the time' and '5' indicated 'all the time'. A mean score was calculated by averaging the scores of the seven questions. A higher score indicated a higher level of well-being.
Change in usage of outdoor exercise facilities | Baseline, Month 1, Month 3
  A self-developed questionnaire will be used to capture the usage of outdoor exercise facilities. Information on the frequency, duration, and types of outdoor exercise facilities used.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Sciences, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JLC, Wong AYL, Ng PHF, Fu SN, Fong KNK, Cheng ASK, Lee KNK, Sun R, Zhang HY, Xiao R. Outdoor Exercise Facility-Based Integrative Mobile Health Intervention to Support Physical Activity, Mental Well-Being, and Exercise Self-Efficacy Among Older Adults With Prefrailty and Frailty in Hong Kong: Pilot Feasibility Randomized Controlled Trial Study. JMIR Mhealth Uhealth. 2025 Jun 5;13:e69259. doi: 10.2196/69259. PMID 40471669